CLINICAL TRIAL: NCT01567228
Title: Delivering Geospatial Intelligence to Health Care Providers
Acronym: CHICA GIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01LM010923-01 (NIH); 1R01LM010923-01 (NIH)
Record Dates: First submitted 2012-01-18; First posted 2012-03-30 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Overweight
Keywords: obesity; overweight; dental caries; school problems; school failure; child BMI > 85th percentile; Needing dental preventive services; Needing academic support for school problems
MeSH Terms: conditions — Overweight; Obesity; Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- routine counseling (control group) (No Intervention): Children will receive typical counseling for obesity prevention, dental caries prevention, or school problems per routine standards for pediatrician anticipatory guidance
- CHICA GIS (Experimental): In randomly assigned experimental clinics, physicians will counsel patients to increase physical activity, seek dental care, or seek academic support services such as tutoring; this counseling will be assisted by an experimental intervention which consist of an electronic medical record that prompts specific counseling in conjunction with a geographic information system. The enhanced electronic medical record will map community resources to support physician counseling and lifestyle modification
  Interventions: Other: CHICA GIS (enhanced electronic medical record)

INTERVENTIONS:
Other: CHICA GIS (enhanced electronic medical record) — An electronic medical record enhanced with geographic information systems will assist physicians in directing patients to community resources for increasing physical activity, preventing dental caries or addressing school problems
  Other Names: CHICA GIS
  Arms: CHICA GIS

SUMMARY:
Physician counseling for physical activity, dental services, and academic support services such as tutoring could be improved through physician knowledge of local community resources and physician counseling directing patients to such services that are near the patient's residential address. This study will test the hypothesis that an electronic medical record enhanced with geographic information systems can improved physician counseling for physical activity, dental services, and academic support services by identifying services that are near the patient's residential address and informing MD's of such info at the point of care.

ELIGIBILITY:
Inclusion Criteria:

* Referrals to three community resources will be studied: dentists (children older than 1 year), after school tutoring services (children older than 7 years), and physical education programs (children older than 5 years).

Exclusion Criteria:

* Inability of parent to complete data collection instruments spoken (via telephone survey) or written in English or Spanish.
* Inability to participate in community based physical activity programs due to health related condition

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1076 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Improved physician counseling | 6 months
  For the intervention clinics, data gathered by CHICA-GIS on the physician worksheet and just-in-time handouts will also allow us to determine the percentage of children who received behavioral counseling about dentistry, school performance, or physical activity by the physician, as well as the percentage of children who were referred to a community resource.

SECONDARY OUTCOMES:
User experience and satisfaction | 24 months
  Surveys will be administered at baseline and end of the trial (18 months) to the entire staff of each practice, in order to document how each practice is organized and provide detailed information about community referral processes. Staff will also be asked about their satisfaction with the CHICA system, CHICA-GIS (Intervention Clinics only), and the community referral module (Intervention Clinics only).

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert C Liu, MD, Principal Investigator — Indiana University
Locations (1):
- Wishard Health Services, Indianapolis, Indiana, United States